CLINICAL TRIAL: NCT03000894
Title: Cognitive Behavioral Therapy for Insomnia as a Transdiagnostic Early Intervention of Mood Disorders: A Randomized Controlled Trial
Brief Title: CBT-I as Early Intervention of Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Kowloon Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chung Ka-Fai, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 16-057
Record Dates: First submitted 2016-12-12; First posted 2016-12-22 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Insomnia Due to Mental Disorder
Keywords: cognitive-behavioral therapy for insomnia; insomnia; mood disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mood Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- CBT-I plus standard care (Experimental): The group CBT-I will receive both CBT-I and standard care. CBT-I covers sleep-wake cycle as well as sleep hygiene education, activity scheduling, stimulus control, sleep restriction, relaxation training, and cognitive therapy. Standard care will include those treatments provided by the psychiatrists according to their clinical needs.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Standard care (No Intervention): Only standard care will be provided to this group. Medications will be prescribed and referral to community nurse, social worker and psychologist will be made by the doctors according to their need.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — This CBT-I is a 4 sessions 60-90 minutes group-based therapy administered by a nurse therapist. Each session has 6-8 participants.
  Arms: CBT-I plus standard care

SUMMARY:
This study aims to investigate the effectiveness of transdiagnostic nurse-administered 4-session group cognitive behavioral therapy for insomnia (CBT-I) plus standard care, compared to standard care alone, for improving sleep and daytime function, enhancing recovery, preventing relapses, and reducing medication burden in patients with the first episode of mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Aged ≥ 18 years
* Able to to communicate in Cantonese and write in Chinese
* First episode of depressive or bipolar disorders according to the DSM-5 diagnostic criteria
* Having received psychiatric treatment for less than 12 months
* Meeting the DSM-5 diagnostic criteria for insomnia disorder for at least 1 month, instead of at least 3 months, as in criterion D.

Exclusion Criteria:

* Significant cognitive impairments and psychotic symptoms, based on a Mini-mental State Examination score of 23 or below and the Positive and Negative Syndrome Scale items on delusions, conceptual disorganization, and hallucinatory behavior at moderate severity or above
* A diagnosis of schizophrenia, delusional disorder, neurocognitive disorders, or learning disability
* Having a highly unstable medical or psychiatric condition (including strong suicidal risk) that requires hospitalization
* Having an untreated sleep disorder, including narcolepsy, obstructive sleep apnea, and periodic leg movement disorder
* Past or current treatment with CBT-I
* Having a fear of speaking in a group setting or refusal to give informed consent
* Refuse to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Chang of subjects'' self-rated score of severity of insomnia symptoms and functional impairment measured by Insomnia Severity Index (ISI) questionnaire | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline

SECONDARY OUTCOMES:
Change of the severity of depression symptoms measured by 17-item Hamilton Depression Rating Scale (HAM-D17) | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of the severity of mania symptoms measured by Young Mania Rating Scale(YMRS) | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of the severity of illness measured by Clinical Global Impressions of Severity (CGI-S) | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of the anxiety and depression state measured by Hospital Anxiety and Depression Scale(HADS) | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' self-rated severity of physical symptoms measured by Somatic Symptom Inventory (SSI) | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' likeliness of dozing measured by Epworth Sleepiness Scale (ESS) | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' self-rated fatigue score measured by Multidimensional Fatigue Inventory (MFI) | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' functioning regarding work/study, social life and family measured by Sheehan Disability Scale (SDS) | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' self-rated score of health state measured by 36-item Short Form Health Survey (SF-36) | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
The number and type of relapses | 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
The number of clinic visits and hospitalizations | 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' perceived stress measured by Perceived Stress Scale | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' sleep-incompatible beliefs and cognition measured by 16-item Dysfunctional Beliefs and Attitudes About Sleep Scale | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' cognitive and somatic arousal prior to sleep onset measured by Pre-sleep Arousal Scale | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' self-efficacy about sleep measured by Self-Efficacy for Sleep Scale | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' sleep inhibitory behavior measured by the Sleep Hygiene Practice Scale | Baseline, 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Change of subjects' credibility to treatment measured by Credibility of treatment rating scale | Baseline and immediate post-treatment, around 8-week post-baseline (CBT-I group), Baseline (Control group)
Prescribed medication burden | 3-month post-baseline, 6-month post-baseline, and 12-month post-baseline
Subjects' satisfaction to CBT-I measured by treatment satisfaction scale | Immediate post-treatment (around 8-week post-baseline)
Subjects' adherence to CBT-I measured by treatment adherence scale | Immediate post-treatment (around 8-week post-baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong